CLINICAL TRIAL: NCT05976217
Title: Safety and Efficacy of Venetoclax in Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, A. Brent Carter, MD, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300010757
Record Dates: First submitted 2023-07-26; First posted 2023-08-04 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: monocyte-derived macrophages; apoptosis resistance
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment (Experimental): Venetoclax 100 mg daily for 3 weeks
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — 100 mg daily by mouth for 3 weeks This drug inhibits a protein (Bcl-2) that protects cells from undergoing programmed cell death.

SUMMARY:
Based on preclinical data, investigators hypothesize that apoptosis resistance in monocyte-derived macrophages (MDMs) have a decisive role in the development of idiopathic pulmonary fibrosis (IPF). Specifically, macrophages from subjects with IPF have increased expression of Bcl-2 in mitochondria. In preclinical models of IPF, a conditional deletion of Bcl-2 in MDMs reverses established fibrosis by inducing apoptosis. Additional evidence to suggest that Bcl-2 expression in MDM mitochondria is a therapeutic target for IPF as administration of the Bcl-2 inhibitor, ABT-199 (Venetoclax), showed marked efficacy in preclinical models of IPF by inducing apoptosis of MDMs and reversing established fibrosis. ABT-199 is an orally available mimetic of the BH3 domain of Bcl-2, which is the domain the anchors Bcl-2 in the mitochondria to inhibit apoptosis. ABT-199 has shown therapeutic efficacy and good safety and tolerability in patients with chronic lymphocytic leukemia. Investigators anticipate that treatment with ABT-199 could result in significant benefit for IPF patients that have a life expectancy of 3-5 years. As there is no curative therapy for IPF, this clinical trial has the potential to substantially alter treatment approaches in patients with IPF.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40-85 years old, male and female.
2. A diagnosis of IPF that fulfills current ATS/ERS Consensus Criteria (1).
3. IPF duration <5 years, based on the date of definitive diagnosis.
4. Ability and willingness to give informed consent and adhere to study requirements.
5. Forced Vital Capacity (FVC) > 50% predicted values.

Exclusion Criteria:

1. Diagnosis of major comorbidities expected to interfere with study participation.
2. History of malignancy within the last 5 years, excluding basal or squamous cell skin cancer.
3. The occurrence of any acute infection requiring systemic antibiotic therapy within 2 weeks prior to Screening (Visit 1).
4. Treatment for >14 days within the preceding month with >20 mg. prednisone (or equivalent) or any treatment during the last month with a cellular immunosuppressant (e.g., cyclophosphamide, methotrexate, calcineurin inhibitors, azathioprine, etc.), given increased risks of opportunistic infections.
5. Concurrent participation in other experimental trials.
6. Fertile women who do not agree to abstinence or an effective form of contraception (as approved by the investigator), or who are breast feeding, for 4 weeks before randomization until 90 days after the last administration of study medication (or placebo).
7. Men who are not surgically sterile and do not agree to remain abstinent from heterosexual intercourse or use effective contraception (as approved by the investigator), and refrain from donating sperm, from the time of giving informed consent until 90 days after the last administration of study medication (or placebo).
8. Subjects with known hypersensitivity to capsule "bulking" agents.
9. A history of bone marrow disorder including aplastic anemia, or marked anemia defined as hemoglobin < 10.0 g/dL (or 6.2 mmol/L).
10. Severe cardiovascular disease, defined as any of the following within the preceding 12 weeks: acute myocardial infarction or unstable angina, a coronary revascularization procedure, congestive heart failure (NYHA Class III or IV), or stroke, including a transient ischemic attack.
11. Evidence of cardiac conducting abnormalities, defined as second- or third-degree AV block not successfully treated with a pacemaker, or a personal or family history of long QT syndrome (QTc interval >450 msec for males or 470 msec for females).
12. End-stage renal disease requiring dialysis.
13. Undergoing transplantation evaluation or listed with the United Network for Organ Sharing (UNOS) as a lung transplantation candidate at the time of enrollment in this trial.
14. Liver function tests (transaminases, alkaline phosphatase, direct and total bilirubin) >2x upper limit of normal values.
15. Systemically administered potent CYP3A4 inhibitors or inducers are prohibited during the 24-week treatment period.

Inhibitors include: pirfenidone, boceprevir, cobicistat, conivaptan, ritonavir, itraconazole, ketoconazole, telaprevir, troleandomycin, voriconazole, clarithromycin, diltiazem, idelalisib, nefazodone, nelfinavir.

Inducers include: carbamazepine, enzalutamide, mitotane, phenytoin, rifampin.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by measuring liver function. | 3 weeks
  complete metabolic panel
Number of participants with treatment-related adverse events as assessed by measuring blood counts. | 3 weeks
  complete blood count

SECONDARY OUTCOMES:
Percentage of monocyte-derived macrophages that undergoing apoptosis. | 3 weeks
  flow cytometry

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - TKC, Birmingham, Alabama
  - UAB, Birmingham, Alabama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Larson-Casey JL, Deshane JS, Ryan AJ, Thannickal VJ, Carter AB. Macrophage Akt1 Kinase-Mediated Mitophagy Modulates Apoptosis Resistance and Pulmonary Fibrosis. Immunity. 2016 Mar 15;44(3):582-596. doi: 10.1016/j.immuni.2016.01.001. Epub 2016 Feb 23. PMID 26921108
- [Result] Larson-Casey JL, Murthy S, Ryan AJ, Carter AB. Modulation of the mevalonate pathway by akt regulates macrophage survival and development of pulmonary fibrosis. J Biol Chem. 2014 Dec 26;289(52):36204-19. doi: 10.1074/jbc.M114.593285. Epub 2014 Nov 5. PMID 25378391
- [Result] Larson-Casey JL, Gu L, Kang J, Dhyani A, Carter AB. NOX4 regulates macrophage apoptosis resistance to induce fibrotic progression. J Biol Chem. 2021 Jul;297(1):100810. doi: 10.1016/j.jbc.2021.100810. Epub 2021 May 21. PMID 34023385
- [Result] Larson-Casey JL, Gu L, Davis D, Cai GQ, Ding Q, He C, Carter AB. Post-translational regulation of PGC-1alpha modulates fibrotic repair. FASEB J. 2021 Jun;35(6):e21675. doi: 10.1096/fj.202100339R. PMID 34038004
- [Result] Gu L, Surolia R, Larson-Casey JL, He C, Davis D, Kang J, Antony VB, Carter AB. Targeting Cpt1a-Bcl-2 interaction modulates apoptosis resistance and fibrotic remodeling. Cell Death Differ. 2022 Jan;29(1):118-132. doi: 10.1038/s41418-021-00840-w. Epub 2021 Aug 20. PMID 34413485